CLINICAL TRIAL: NCT03356704
Title: Is the Combined Plexus Block a Real Alternative for Hip Fracture Surgery in the Elderly? A Comparison With General Anesthesia and Continuous Spinal Anesthesia Using a Propensity Score in a Retrospective Cohort Study.
Brief Title: Combined Plexus Block for Hip Fracture Surgery.
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0229
Record Dates: First submitted 2017-10-26; First posted 2017-11-29 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-10

CONDITIONS: Hip Fractures
Keywords: adults
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General anaesthesia: Patient who had surgery for femoral neck fracture from January 2014 to December 2016 and had general anesthesia
  Interventions: Other: no intervention
- continued spinal anesthesia: Patient who had surgery for femoral neck fracture from January 2014 to December 2016 and had continued spinal anesthesia
  Interventions: Other: no intervention
- peripheral nerve blocks: Patient who had surgery for femoral neck fracture from January 2014 to December 2016 and had peripheral nerve blocks
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Observational study

SUMMARY:
Hip fracture surgery requires high risk anesthetic procedure for elderly patients (1). General anesthesia, continuous spinal anesthesia and peripheral nerve blocks are three anesthetic techniques possible. Continuous spinal anesthesia has proven its efficacity to provide an intraoperative haemodynamic stability wich guarantees good patients outcomes (2), in comparison with general anesthesia but there is poor evidence in the literature concerning the use of peripheral nerve blocks.

The primary objective of this study was to compare intraoperative haemodynamic stability provides by peripheral nerve block versus general anesthesia and continuous spinal anesthesia.

Secondary outcomes included : use of vasoactive drugs, opioids consumption, lengh of stay and inhospital mortality.

DETAILED DESCRIPTION:
After receiving the ethic approval from the "CERAR", the investigators retrospectively identified all patients who underwent hip fracture surgery from January 1 2015, to December 31, 2016 in the CHU of Montpellier. The exclusion criteria were: multiple trauma victims, two hip fractures in the same patient and single shot spinal anesthesia. In our institution the investigators used to perform three types of anesthesia: general anesthesia (GA), continuous spinal anesthesia (CSA) and combined plexus blocks (CPB). The investigators therefore made three groups GA, CSA and CPB and used a propensity score to make these groups comparable. The matching criteria were age, arterial hypertension, ASA status, Frailty score, chronic cardiac failure and type of surgery.

ELIGIBILITY:
Inclusion criteria:

* Adult
* Hip fracture surgery

Exclusion criteria:

* Multiple trauma victims
* Second hip fracture in same patient
* Single shot spinal anesthesia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adults patients operated for hip fracture between 1 January 2015 and 31 December 2016.
Sampling Method: Probability Sample
Enrollment: 593 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Intraoperative hypotension | 1 day
  Decrease of at least 30% of mean arterial pressure

SECONDARY OUTCOMES:
measure the total consumption of the vasopressive molecules | 1 day
  measure the total consumption of the vasopressive molecules (necessary when the voltage drops by more than 30% compared to the average reference voltage) : Use of vasoactive drugs
Length of stay | 1 day
  Length of stay
compare the use of emergency antalgics | 1 day
  compare the use of emergency antalgics : opioids consumption
Inhospital mortality | 1 day
  Inhospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Capdevila, MD, PhD, Study Director — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Mounet B, Choquet O, Swisser F, Biboulet P, Bernard N, Bringuier S, Capdevila X. Impact of multiple nerves blocks anaesthesia on intraoperative hypotension and mortality in hip fracture surgery intermediate-risk elderly patients: A propensity score-matched comparison with spinal and general anaesthesia. Anaesth Crit Care Pain Med. 2021 Aug;40(4):100924. doi: 10.1016/j.accpm.2021.100924. Epub 2021 Jul 1. PMID 34217841